CLINICAL TRIAL: NCT06327620
Title: A Novel Alternative Treatment Of Oral Lichen Planus
Brief Title: Treatment Of Oral Lichen Planus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Wafaa Saleh, Assistant professor, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: A002021015
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Lichen Planus
Keywords: lichen planus; Treatment
MeSH Terms: conditions — Lichen Planus | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daivobet Ointment (Experimental): Daivobet Ointment Arm: Patients in this arm will be asked to topically apply Daivobet ointment three times daily for four weeks
  Interventions: Combination Product: Daivobet ointment, topical steroids
- Topical steroids (Active Comparator): Patients in this arm will be asked to topically apply a steroid ointment three times daily for four weeks.
  Interventions: Combination Product: Daivobet ointment, topical steroids

INTERVENTIONS:
Combination Product: Daivobet ointment, topical steroids — Daivobet Ointment: This intervention involves the topical application of Daivobet ointment, which is a combination of calcipotriol and betamethasone. The application is to be done three times daily for four weeks.
  Topical Steroid: This intervention entails the topical application of a steroid ointment three times daily for four weeks. The specific steroid and its details are not disclosed in the provided information.

SUMMARY:
This novel project aims to explore an alternative treatment for oral lichen planus (OLP), a challenging condition with limited therapeutic options. The proposed treatment involves the topical application of Daivobet ointment, a combination of calcipotriol (vitamin D analog) and betamethasone (corticosteroid), which has shown promising results in the treatment of psoriasis Vulgaris.

The study will involve 15 patients aged 30-60 years with clinically confirmed intra-oral erosive lichen planus, some of whom have not responded to current therapies. Participants will apply Daivobet ointment three times daily for four weeks, with clinical assessments conducted at the beginning, and at the end of the second and fourth weeks.

Inclusion criteria require the presence of bilateral oral erosive lichen planus lesions, with clinical and histopathological confirmation based on the World Health Organization's modified definition. Exclusion criteria include histological signs of dysplasia, use of drugs possibly causing lichenoid reactions, recent treatment for OLP, and hypersensitivity to the study drug.

Clinical evaluations will employ a scoring system based on lesion characteristics, including ulceration, erythema, and reticulation, measured with a calibrated grid. Subjective responses will be assessed through discomfort scores on a visual analog scale, and a questionnaire will capture any adverse effects. Digital photographs will document visual changes, and incisional biopsies will be performed to confirm the diagnosis.

The project aims to provide valuable insights into the efficacy and safety of the Daivobet ointment as a potential alternative treatment for oral lichen planus, offering hope for improved outcomes for patients suffering from this challenging condition.

DETAILED DESCRIPTION:
This clinical study aims to explore a novel alternative treatment for oral lichen planus (OLP) utilizing Daivobet ointment, a combination of calcipotriol and betamethasone. The protocol is designed to provide in-depth technical information on patient selection, treatment procedures, clinical assessments, and statistical analyses, ensuring a comprehensive understanding of the study's methodology.

Patient Selection:

Fifteen patients aged 30-60 with bilateral intra-oral erosive lichen planus symptoms will be recruited from the department of Oral Medicine and Diagnosis at the Faculty of Dentistry, Kafr Elsheikh University. Participants with a history of unresponsiveness to current therapies will undergo histopathological confirmation through incisional biopsy.

Inclusion Criteria:

Presence of bilateral oral erosive lichen planus lesions. Clinical and histopathological diagnosis of oral lichen planus based on a modified definition of the World Health Organization (WHO).

Exclusion Criteria:

Histological signs of dysplasia. Use of drugs possibly causing a lichenoid reaction and lesions in contact with dental amalgam restorations.

Any topical or systemic medications used in the treatment of oral lichen planus within four weeks before the study.

Patients with a history of hypersensitivity to the drug used in the current study.

Clinical Assessment:

Patients will be instructed to topically apply Daivobet ointment on one side and a topical steroid on the other side three times daily for four weeks. Clinical evaluations will be conducted at the study's onset, with baseline parameters recorded, and reassessed at the end of the second and fourth weeks.

Objective Response:

Lesions of oral lichen planus will be scored using a scaled tongue blade, categorizing them from 0 (no lesion) to 5 (erosive area >1cm2). Quantitative measurements will be calculated using a transparent grid to obtain the total area of the lesion.

Subjective Response:

Discomfort scores will be recorded on a visual analog scale ranging from 0 to 3, and a questionnaire documenting potential adverse effects will be completed. Patients will rank the severity of their discomfort.

Biopsy Specimens and Laboratory Investigations:

Incisional biopsy specimens will be obtained under local anesthesia, incorporating both clinically normal and diseased tissues. The specimens will undergo routine histologic study, confirming the diagnosis through formalin-fixed, paraffin-embedded, hematoxylin-and eosin-stained sections.

Statistical Analysis:

Data analysis will be performed using SPSS version 16 for Windows. The normality of data will be assessed using Shapiro-Wilk tests. Descriptive statistics, median, minimum, and maximum tests will be employed to describe the measure of central tendency and dispersion in each group. Groups will be compared using the Mann-Whitney U test. For non-parametric continuous variables, the degree of improvement will be calculated, and the mean value for the degree of improvement used to compare between groups. The significance level will be set at P ≤ 0.05.

Patient Registry Procedures:

Quality assurance plan addressing data validation, registry procedures, site monitoring, and auditing.

Data checks to compare entered data against predefined rules for range or consistency.

Source data verification assessing the accuracy, completeness, or representativeness of registry data by comparing it to external sources.

Data dictionary containing detailed descriptions of each variable, including source, coding information, and normal ranges.

Standard Operating Procedures covering registry operations and analysis activities, including patient recruitment, data collection, management, analysis, reporting for adverse events, and change management.

Sample size assessment specifying the number of participants or participant years necessary to demonstrate an effect.

Plan for missing data addressing situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing due to data inconsistency or out-of-range results.

Statistical analysis plan describing the analytical principles and techniques employed to address the primary and secondary objectives, as specified in the study protocol or plan.

ELIGIBILITY:
Inclusion Criteria:

Age between 30-60 years. Clinical signs and symptoms of bilateral intra-oral erosive lichen planus. History of unresponsiveness to currently available therapy. Histopathological confirmation by incisional biopsy. Willingness to topically apply Daivobet ointment in one side and topical steroid in the other side three times daily for 4 weeks.

Exclusion Criteria:

* Histological signs of dysplasia. Use of drugs possibly causing a lichenoid reaction. Lesions in contact with dental amalgam restorations. Any topical or systemic medications used in the treatment of oral lichen planus within four weeks before the study.

History of hypersensitivity to the drug used in the current study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement of Oral Lichen Planus Lesions | End of the second and fourth weeks of treatment.
  Assessment of the degree of clinical improvement based on the reduction in the severity of oral lichen planus lesions.

SECONDARY OUTCOMES:
Objective Response Score | End of the second and fourth weeks of treatment
  Measurement of the objective response using a scaled tongue blade to score oral lichen planus lesions based on defined criteria.
Subjective Response Score | Start of the study and at the end of the second and fourth weeks of treatment.
  Evaluation of subjective response through discomfort scores recorded on a visual analog scale, ranking the severity of discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No